CLINICAL TRIAL: NCT04639765
Title: Responses to Information on Treatments for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel R. Strunk, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020B0259
Record Dates: First submitted 2020-11-11; First posted 2020-11-20 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Depressive Symptoms
Keywords: depression; treatment preference; treatment information
MeSH Terms: conditions — Depression | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- No video (No Intervention): This condition involves no video presentation.
- CBT without Personalization (Experimental): Video provides information about cognitive behavioral therapy.
  Interventions: Other: CBT without Personalization
- CBT with Personalization (Experimental): Video provides information about cognitive behavioral therapy and describes how treatment can be personalized.
  Interventions: Other: CBT with Personalization
- ADM without Personalization (Experimental): Video provides information about antidepressant medications.
  Interventions: Other: ADM without Personalization
- ADM with Personalization (Experimental): Video provides information about antidepressant medications and describes how treatment can be personalized.
  Interventions: Other: ADM with Personalization
- Combined Treatment without Personalization (Experimental): Video provides information on the combined treatment of cognitive behavioral therapy with antidepressant medications.
  Interventions: Other: Combined Treatment without Personalization
- Combined Treatment with Personalization (Experimental): Video provides information on the combined treatment of cognitive behavioral therapy with antidepressant medications and describes how treatment can be personalized.
  Interventions: Other: Combined Treatment with Personalization

INTERVENTIONS:
Other: CBT without Personalization — Intervention involves a video describing CBT without a message about personalization.
  Arms: CBT without Personalization
Other: CBT with Personalization — Intervention involves a video describing CBT with a message about personalization.
  Arms: CBT with Personalization
Other: ADM without Personalization — Intervention involves a video describing antidepressant medication without a message about personalization.
  Arms: ADM without Personalization
Other: ADM with Personalization — Intervention involves a video describing antidepressant medication with a message about personalization.
  Arms: ADM with Personalization
Other: Combined Treatment without Personalization — Intervention involves a video describing the combination of cognitive behavior therapy and antidepressant medication without a message about personalization.
  Arms: Combined Treatment without Personalization
Other: Combined Treatment with Personalization — Intervention involves a video describing the combination of cognitive behavior therapy and antidepressant medication with a message about personalization.
  Arms: Combined Treatment with Personalization

SUMMARY:
The purpose of this study is to determine the impact of different messages about depression treatments.

DETAILED DESCRIPTION:
Participants recruited through Amazon Mechanical Turk (MTurk) will complete a screening questionnaire and provided the opportunity to consent to participate. Upon entry to the study, eligible participants will complete several questionnaires pre- and post-randomization. Randomization will be to view either a video detailing a type of depression treatment (cognitive behavioral therapy, antidepressant medication, or the combination of both treatments) with and without an emphasis on personalization. A no video condition is also included.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 Score indicating a history of elevated depression symptoms
* A high MTurk completion rate
* Must pass all attention checks inserted into the questionnaires
* No history of treatment for depression

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Regressed change from baseline in expectations on the Credibility/Expectancy Questionnaire (CEQ) | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  The CEQ is a validated, commonly used measure assessing views of the credibility and expectations for benefit from a treatment.
Regressed change from baseline in prognostic pessimism on an adapted version of the Perceptions of Depression Scale (PDS) | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  Measured using an adapted version of the PDS, a validated scale measuring general prognostic pessimism. Minor changes to wording were made to directly address the three different interventions in the study (CBT, ADM, Combined Treatment).

SECONDARY OUTCOMES:
Regressed change from baseline in affect on the Positive and Negative Affectivity Scale (PANAS) | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  The PANAS is a widely used measure for positive and negative affect, and has been shown to be valid and reliable.
Regressed Change from baseline on the Beck Hopelessness Scale (BHS) | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  The BHS is the most widely used measure for hopelessness, and has been shown to be valid and reliable.
Regressed change from baseline in personal and perceived depression stigma on the Depression Stigma Scale (DSS). | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  The DSS is a valid and reliable measure for assessing personal and perceived stigma related to depression. The scale contains two subscales: personal stigma and perceived stigma.
Regressed change from baseline in beliefs on the etiology of depression on the Reasons for Depression Questionnaire (RFD). | Up to 90 minutes to complete assessment. Assessed immediately pre- and post-intervention (on the same day)
  The RFD is a valid and reliable measure for assessing one's beliefs on the etiology of depression.
Willingness to take a next step. | Up to 90 minutes to complete assessment. Assessed at the end of the study questionnaires (same day)
  Participants are given the option to learn more about finding cognitive behavioral therapy, antidepressant medications, or combination therapy. Based on their responses, they are provided links to relevant websites. This approach has been adopted from traditional marketing research to assess participants' responsiveness to a message.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Strunk, PhD, Principal Investigator — Professor
Locations (1):
- Psychology Building 1835 Neil Avenue, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified data upon reasonable request.
Time Frame: Data available for two years post-publication or at the end of the project if no papers are published.
Access Criteria: Will share de-identified data upon reasonable request.